CLINICAL TRIAL: NCT02100722
Title: Fractional Flow Reserve Versus Angiography for Multivessel Evaluation (FAME) 3 Trial A Comparison of Fractional Flow Reserve-Guided Percutaneous Coronary Intervention and Coronary Artery Bypass Graft Surgery in Patients With Multivessel Coronary Artery Disease
Brief Title: A Comparison of Fractional Flow Reserve-Guided Percutaneous Coronary Intervention and Coronary Artery Bypass Graft Surgery in Patients With Multivessel Coronary Artery Disease
Acronym: FAME 3
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: VZW Cardiovascular Research Center Aalst (Other); Catharina Ziekenhuis Eindhoven (Other); Golden Jubilee National Hospital (Other Government); University of California, Irvine (Other); Medtronic (Industry); Abbott Medical Devices (Industry); Genae (Industry); King's College Hospital NHS Trust (Other); Houston Methodist DeBakey Heart & Vascular Center (Other)
Responsible Party: Principal Investigator, William Fearon, Principle Investigator, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FAME 3
Record Dates: First submitted 2014-03-21; First posted 2014-04-01 (Estimated); Results first posted 2022-01-20 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Coronary Disease; Coronary Stenosis
MeSH Terms: conditions — Coronary Disease; Coronary Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FFR guided PCI (Active Comparator): Patients undergoing PCI will have FFR measured with a St. Jude Medical coronary pressure wire across all lesions. If the FFR is ≤0.80, then PCI will be performed with the Medtronic Resolute Integrity (or Onyx) drug-eluting stent (DES) as per usual routine. If the FFR is >0.80 then PCI will be deferred. Only those sites with prior experience measuring FFR will be included in the FAME 3 trial. These patients in whom FFR of a particular lesion was not possible will be included in all analyses based on the intention to treat principle.
  Interventions: Procedure: FFR guided PCI; Device: Resolute Integrity Stent; Device: Resolute Onyx Stent
- CABG (Active Comparator): CABG will be performed as per clinical routine at each participating center. Both off-pump and on-pump surgery are acceptable, as long as the surgeon and the site are experienced in the particular technique. An internal mammary graft to the LAD should be attempted in all cases, if feasible. Complete arterial revascularization is strongly recommended, however, each center should use a conduit strategy with which they are most comfortable. All vessels ≥ 1,5 mm in diameter and with ≥ 50% stenosis should be bypassed, if technically feasible.
  Interventions: Procedure: CABG

INTERVENTIONS:
Procedure: FFR guided PCI
  Other Names: Fractional Flow Reserve-Guided PCI
  Arms: FFR guided PCI
Procedure: CABG — Coronary Artery Bypass Graft Surgery (CABG)
  Arms: CABG
Device: Resolute Integrity Stent — Durable polymer zotarolimus-eluting stent
  Arms: FFR guided PCI
Device: Resolute Onyx Stent — Durable polymer zotarolimus-eluting stent
  Arms: FFR guided PCI

SUMMARY:
The purpose of this study is to determine whether Fractional flow reserve (FFR, (coronary pressure wire-based index for assessing the ischemic potential of a coronary lesion)-guided percutaneous coronary intervention (PCI) in patients with multivessel coronary artery disease (CAD) will result in similar outcomes to coronary artery bypass graft surgery (CABG).

DETAILED DESCRIPTION:
The FAME 3 trial is a multicenter, international, randomized, controlled noninferiority trial. All patients with multivessel CAD (not involving the left main) will be screened by the site's Heart Team (including but not limited to an interventional cardiologist, cardiac surgeon and research coordinator). If all agree that the patient can be treated either with FFR-guided PCI or CABG, and all inclusion criteria are met and no exclusion criteria are met, then the patient will be randomized.

Baseline clinical, functional, laboratory and electrocardiographic data will be obtained. Patients will receive treatment within 4 weeks of randomization. Patients randomized to CABG will receive state of the art therapy at the discretion of the local surgeon with a strong emphasis on arterial revascularization. Patients undergoing PCI will have FFR measured with a St. Jude Medical coronary pressure wire across all lesions. If the FFR is ≤0.80, then PCI will be performed with the Medtronic Resolute Integrity drug-eluting stent (DES) as per usual routine. If the FFR is >0.80 then PCI will be deferred.

All patients will receive medical therapy as per published guidelines. Patients will follow-up at 1 and 6 months, and 1 and 3 years with an evaluation of clinical status, functional status, medications and events. Follow-up may be extended to 5 years, if funding allows.

Core lab analyses will include formal quantitative coronary angiography (QCA) of the baseline angiograms with calculation of the Synergy between Percutaneous Coronary Intervention with Taxus and Cardiac Surgery (SYNTAX) score and Functional SYNTAX Score.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age ≥ 21 years with angina and/or evidence of myocardial ischemia
* 2. Three vessel CAD, defined as ≥ 50% diameter stenosis by visual estimation in each of the three major epicardial vessels or major side branches, but not involving left main coronary artery, and amenable to revascularization by both PCI and CABG as determined by the Heart Team. Patients with a non-dominant right coronary artery may be included if only the left anterior descending artery (LAD) and left circumflex have ≥50% stenosis
* 3. Willing and able to provide informed, written consent

Exclusion Criteria:

* 1. Requirement for other cardiac or non-cardiac surgical procedure (e.g., valve replacement, carotid revascularization)
* 2. Cardiogenic shock and/or need for mechanical/pharmacologic hemodynamic support
* 3. Recent STEMI (<5 days prior to randomization)
* 4. Ongoing Non STEMI with biomarkers (cardiac troponin) still rising
* 5. Known left ventricular ejection fraction <30%
* 6. Life expectancy < 2 years
* 7. Requiring renal replacement therapy
* 8. Undergoing evaluation for organ transplantation
* 9. Participation or planned participation in another clinical trial, except for observational registries
* 10. Pregnancy
* 11. Inability to take dual antiplatelet therapy for six months
* 12. Previous CABG
* 13. Left main disease requiring revascularization
* 14. Extremely calcified or tortuous vessels precluding FFR measurement
* 15. Any target lesion with in-stent drug-eluting stent restenosis

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Actual)
Dates: Start 2014-08-25 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2025-04 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: William F Fearon, MD, Study Chair — Stanford University; Nico HJ Pijls, MD, PhD, Principal Investigator — Catharina Hospital Eindhoven, The Netherlands; Bernard De Bruyne, MD, PhD, Principal Investigator — VZW Cardiovascular Research Center Aalst
Locations (46):
- United States (13):
  - Palo Alto VA, Palo Alto, California
  - Stanford University, Stanford, California
  - Atlanta VA Medical Center, Decatur, Georgia
  - Jesse Brown VA Medical Center, Chicago, Illinois
  - University of Kansas Medical Center, Lawrence, Kansas
  - Lexinton VA, Lexington, Kentucky
  - University of Kentucky Medical Center, Lexington, Kentucky
  - Baystate Medical Center, Springfield, Massachusetts
  - HealthEast St. Joseph's Hospital, Saint Paul, Minnesota
  - Penn Presbyterian Medical Center, Philadelphia, Pennsylvania
  - Centennial Heart, Nashville, Tennessee
  - Houston Methodist Hospital, Houston, Texas
  - University of Virginia, Charlottesville, Virginia
- Australia (5):
  - Peninsula Health, Frankston
  - St. Vincent's Hospital Melbourne, Melbourne
  - Concord Hospital, Sydney
  - Royal North Shore, Sydney
  - University of Sydney, Sydney
- Cardiovascular Center Aalst, Aalst, Belgium
- Canada (3):
  - Le'Centre Hospitalier de l'Universite de Montreal, Montreal
  - York PCI Group INC, Ontario
  - University of Ottawa Heart Institute, Ottawa
- Masaryk University and University Hospital Brno, Brno, Czechia
- Rigshospitalet University Hospital, Copenhagen, Denmark
- Cardiovascular Hospital, Lyon, France
- Hungarian Institute of Cardiology, Budapest, Hungary
- Vilnius University Hospital Santariskiu Klinikos, Vilnius, Lithuania
- Netherlands (3):
  - Catharina Hospital Eindhoven, Eindhoven
  - HagaZiekenhuis, The Hague
  - Isala Klinieken, Zwolle
- Waikato Hospital, Hamilton, New Zealand
- Stavanger University Hospital, Stavanger, Norway
- Serbia (2):
  - University Clinical Center of Serbia, Belgrade
  - Clinical Center Kragujevac, Kragujevac
- Asan Medical Center, Seoul, South Korea
- Sweden (3):
  - Sahlgrenska University Hospital, Gothenburg
  - Danderyds Sjukhus, Stockholm
  - Karolinska Institutet, Dep of clinical science and education, Södersjukhuset, Stockholm
- United Kingdom (8):
  - Wales Heart Research Institute, Cardiff
  - University Hospitals Coventry and Warwickshire, Coventry and Warwickshire
  - Golden Jubilee National Hospital, Glasgow
  - Kings College Hospital, London
  - St. Thomas' Hospital, London
  - Wythenshawe Hospital, Manchester
  - Oxford University Hospital NHS Trust, Oxford
  - Southampton University Hospitals NHS Trust, Southhampton

REFERENCES:
- [Background] Zimmermann FM, De Bruyne B, Pijls NH, Desai M, Oldroyd KG, Park SJ, Reardon MJ, Wendler O, Woo J, Yeung AC, Fearon WF. Rationale and design of the Fractional Flow Reserve versus Angiography for Multivessel Evaluation (FAME) 3 Trial: a comparison of fractional flow reserve-guided percutaneous coronary intervention and coronary artery bypass graft surgery in patients with multivessel coronary artery disease. Am Heart J. 2015 Oct;170(4):619-626.e2. doi: 10.1016/j.ahj.2015.06.024. Epub 2015 Jul 9. PMID 26386784
- [Background] Zimmermann FM, De Bruyne B, Pijls NHJ, Desai M, Oldroyd KG, Reardon MJ, Wendler O, Woo J, Yeung AC, Fearon WF. A protocol update of the Fractional Flow Reserve versus Angiography for Multivessel Evaluation (FAME) 3 trial: A comparison of fractional flow reserve-guided percutaneous coronary intervention and coronary artery bypass graft surgery in patients with multivessel coronary artery disease. Am Heart J. 2019 Aug;214:156-157. doi: 10.1016/j.ahj.2019.04.012. Epub 2019 Apr 29. No abstract available. PMID 31207442
- [Result] Fearon WF, Zimmermann FM, De Bruyne B, Piroth Z, van Straten AHM, Szekely L, Davidavicius G, Kalinauskas G, Mansour S, Kharbanda R, Ostlund-Papadogeorgos N, Aminian A, Oldroyd KG, Al-Attar N, Jagic N, Dambrink JE, Kala P, Angeras O, MacCarthy P, Wendler O, Casselman F, Witt N, Mavromatis K, Miner SES, Sarma J, Engstrom T, Christiansen EH, Tonino PAL, Reardon MJ, Lu D, Ding VY, Kobayashi Y, Hlatky MA, Mahaffey KW, Desai M, Woo YJ, Yeung AC, Pijls NHJ; FAME 3 Investigators. Fractional Flow Reserve-Guided PCI as Compared with Coronary Bypass Surgery. N Engl J Med. 2022 Jan 13;386(2):128-137. doi: 10.1056/NEJMoa2112299. Epub 2021 Nov 4. PMID 34735046
- [Derived] Takahashi K, Otsuki H, Zimmermann FM, Ding VY, Piroth Z, Oldroyd KG, Wendler O, Reardon MJ, Desai M, Woo YJ, Yeung AC, De Bruyne B, Pijls NHJ, Fearon WF; FAME 3 Trial Investigators. Outcomes After CABG Compared With FFR-Guided PCI in Patients Presenting With Acute Coronary Syndrome. JACC Cardiovasc Interv. 2025 Apr 14;18(7):838-848. doi: 10.1016/j.jcin.2025.01.434. PMID 40240081
- [Derived] Fearon WF, Zimmermann FM, Ding VY, Takahashi K, Piroth Z, van Straten AHM, Szekely L, Davidavicius G, Kalinauskas G, Mansour S, Kharbanda R, Ostlund-Papadogeorgos N, Aminian A, Oldroyd KG, Al-Attar N, Jagic N, Dambrink JE, Kala P, Angeras O, MacCarthy P, Wendler O, Casselman F, Witt N, Mavromatis K, Miner SES, Sarma J, Engstrom T, Christiansen EH, Tonino PAL, Reardon MJ, Otsuki H, Kobayashi Y, Hlatky MA, Mahaffey KW, Desai M, Woo YJ, Yeung AC, Pijls NHJ, De Bruyne B. Outcomes after fractional flow reserve-guided percutaneous coronary intervention versus coronary artery bypass grafting (FAME 3): 5-year follow-up of a multicentre, open-label, randomised trial. Lancet. 2025 Apr 26;405(10488):1481-1490. doi: 10.1016/S0140-6736(25)00505-7. Epub 2025 Mar 30. PMID 40174598
- [Derived] Takahashi K, Otsuki H, Zimmermann FM, Ding VY, Engstrom T, Horsted Thyregod HG, Beleslin B, Putnik S, Tapp L, Barker T, Redwood S, Young C, Bech GJ, Hoohenkerk GJF, De Bruyne B, Pijls NHJ, Fearon WF; FAME 3 Trial Investigators. FFR-Guided Percutaneous Coronary Intervention vs Coronary Artery Bypass Grafting in Patients With Diabetes. JAMA Cardiol. 2025 Jun 1;10(6):603-608. doi: 10.1001/jamacardio.2025.0095. PMID 40072460
- [Derived] Takahashi K, Otsuki H, Zimmermann FM, Ding VY, Oldroyd KG, Wendler O, Reardon MJ, Woo YJ, Yeung AC, Pijls NHJ, De Bruyne B, Fearon WF; FAME 3 Trial Investigators. Sex Differences in Patients Undergoing FFR-Guided PCI or CABG in the FAME 3 Trial. JACC Cardiovasc Interv. 2025 Jan 27;18(2):157-167. doi: 10.1016/j.jcin.2024.09.030. Epub 2024 Dec 4. PMID 39641725
- [Derived] Otsuki H, Takahashi K, Zimmermann FM, Mavromatis K, Aminian A, Jagic N, Dambrink JE, Kala P, MacCarthy P, Witt N, Kobayashi Y, Takahashi T, Woo YJ, Yeung AC, De Bruyne B, Pijls NHJ, Fearon WF; FAME 3 Trial Investigators. Impact of a Chronic Total Occlusion on Outcomes After FFR-Guided PCI or Coronary Bypass Surgery: A FAME 3 Substudy. Circ Cardiovasc Interv. 2024 Nov;17(11):e014300. doi: 10.1161/CIRCINTERVENTIONS.124.014300. Epub 2024 Nov 6. PMID 39502029
- [Derived] Zimmermann FM, Ding VY, Pijls NHJ, Piroth Z, van Straten AHM, Szekely L, Davidavicius G, Kalinauskas G, Mansour S, Kharbanda R, Ostlund-Papadogeorgos N, Aminian A, Oldroyd KG, Al-Attar N, Jagic N, Dambrink JE, Kala P, Angeras O, MacCarthy P, Wendler O, Casselman F, Witt N, Mavromatis K, Miner SES, Sarma J, Engstrom T, Christiansen EH, Tonino PAL, Reardon MJ, Otsuki H, Kobayashi Y, Hlatky MA, Mahaffey KW, Desai M, Woo YJ, Yeung AC, De Bruyne B, Fearon WF; FAME 3 Investigators. Fractional Flow Reserve-Guided PCI or Coronary Bypass Surgery for 3-Vessel Coronary Artery Disease: 3-Year Follow-Up of the FAME 3 Trial. Circulation. 2023 Sep 19;148(12):950-958. doi: 10.1161/CIRCULATIONAHA.123.065770. Epub 2023 Aug 21. PMID 37602376
- [Derived] Piroth Z, Otsuki H, Zimmermann FM, Ferenci T, Keulards DCJ, Yeung AC, Pijls NHJ, De Bruyne B, Fearon WF. Prognostic Value of Measuring Fractional Flow Reserve After Percutaneous Coronary Intervention in Patients With Complex Coronary Artery Disease: Insights From the FAME 3 Trial. Circ Cardiovasc Interv. 2022 Nov;15(11):884-891. doi: 10.1161/CIRCINTERVENTIONS.122.012542. Epub 2022 Sep 19. PMID 36121706
- [Derived] Fearon WF, Zimmermann FM, Ding VY, Zelis JM, Piroth Z, Davidavicius G, Mansour S, Kharbanda R, Ostlund-Papadogeorgos N, Oldroyd KG, Wendler O, Reardon MJ, Woo YJ, Yeung AC, Pijls NHJ, De Bruyne B, Desai M, Hlatky MA; FAME 3 Investigators. Quality of Life After Fractional Flow Reserve-Guided PCI Compared With Coronary Bypass Surgery. Circulation. 2022 May 31;145(22):1655-1662. doi: 10.1161/CIRCULATIONAHA.122.060049. Epub 2022 Apr 2. PMID 35369704
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/26386784

RESULTS

PARTICIPANT FLOW:
Groups:
- FFR Guided PCI: Patients undergoing Percutaneous Coronary Intervention (PCI) will have Fractional Flow Reserve (FFR) measured with a St. Jude Medical coronary pressure wire across all lesions. If the FFR is ≤0.80, then PCI will be performed with the Medtronic Resolute Integrity (or Onyx) drug-eluting stent as per usual routine.
- CABG: Coronary-artery bypass grafting (CABG) performed per clinical routine (both off-pump and on-pump surgery acceptable).
Period: Overall Study
Arm/Group | FFR Guided PCI | CABG
Started | 757 | 743
Underwent Alternate Procedure (Due to patient/physician refusal to undergo/perform procedure or an acute event leading to an alternative treatment) | 11 | 37
Completed | 0 | 0
Not Completed | 757 | 743
Not completed — Withdrawal pre-procedure | 4 | 9
Not completed — Withdrawal post-procedure | 0 | 3
Not completed — Lost to Follow-up | 2 | 2
Not completed — Continuing on study | 751 | 729

BASELINE CHARACTERISTICS:
Groups:
- FFR Guided PCI: Patients undergoing PCI with measured FFR ≤0.80 have PCI performed with Medtronic Resolute Integrity (or Onyx) drug-eluting stent.
- CABG: CABG performed per clinical routine (both off-pump and on-pump surgery acceptable).
- Total: Total of all reporting groups
Arm/Group | FFR Guided PCI | CABG | Total
Number analyzed (Participants) | 757 | 743 | 1500
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.2 (8.6) | 65.1 (8.3) | 65.2 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 141 | 124 | 265
  Male | 616 | 619 | 1235
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 711 | 686 | 1397
  Non-white | 46 | 57 | 103
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 28.6 (4.5) | 28.7 (4.3) | 28.7 (4.4)
Diabetes [Count of Participants; unit: Participants]
  Overall | 214 | 214 | 428
  Insulin-dependent | 55 | 61 | 116
  Non-insulin-dependent | 159 | 153 | 312
Hypertension [Count of Participants; unit: Participants] | 538 | 556 | 1094
Smoking Status [Count of Participants; unit: Participants]
  Current tobacco user | 145 | 136 | 281
  Previous tobacco user | 296 | 296 | 592
Family history of coronary artery disease [Count of Participants; unit: Participants] | 246 | 213 | 459
Previous myocardial infarction [Count of Participants; unit: Participants] | 252 | 248 | 500
Previous PCI [Count of Participants; unit: Participants] | 98 | 104 | 202
History of transient ischemic attack (TIA) or cerebral vascular accident (CVA) [Count of Participants; unit: Participants] | 49 | 56 | 105
Kidney disease [Count of Participants; unit: Participants] | 37 | 44 | 81
Noninvasive test for ischemia [Count of Participants; unit: Participants] | 311 | 301 | 612
Left ventricular ejection fraction (LVEF) ≤50% [Count of Participants; unit: Participants] | 137 | 130 | 267
Hospitalized with Non-ST elevation-acute coronary syndrome (NSTE-ACS) [Count of Participants; unit: Participants] | 300 | 287 | 587

OUTCOME MEASURES:

1. Primary Outcome: MACCE
Description: Death, MI, stroke and any repeat revascularization (MACCE) will be evaluated at 1 year, where subjects contribute data from time of randomization until the occurrence of MACCE or one year follow-up, whichever occurs first. Subjects who die or are lost to follow up before 1 year will be censored at their last recorded activity.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | FFR Guided PCI | CABG
Number analyzed (Participants) | 757 | 743
Participants | 80 | 51
Statistical Analysis 1: Comparison: FFR Guided PCI vs CABG; A sample of 712 patients per group (1424 for the entire trial) would be required in order to achieve 90% power to claim noninferiority; Test type: Non-Inferiority — Noninferiority of FFR-guided PCI to CABG was prespecified as an upper boundary of less than 1.65 for the 95% confidence interval of the hazard ratio; p = 0.35, Regression, Cox; Hazard Ratio (HR) = 1.5, 95% CI 2-sided [1.1 to 2.2]

2. Secondary Outcome: Key Secondary Outcome: Composite of Death From Any Cause, Myocardial Infarction, or Stroke
Description: Death, MI, or stroke at 3-year follow-up
Time Frame: 3 years
Population: FFR-guided PCI vs CABG
Measure: Count of Participants; unit: Participants
Groups:
- CABG: CABG
Arm/Group | FFR Guided PCI | CABG
Number analyzed (Participants) | 757 | 743
Participants | 91 | 68

3. Secondary Outcome: Number of Participants Experiencing Death, MI, or Stroke
Description: Subjects who died or are lost to follow up before this time were censored at their last recorded activity.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | FFR Guided PCI | CABG
Number analyzed (Participants) | 757 | 743
Participants | 55 | 39

4. Secondary Outcome: Death
Description: Death evaluated excluding patients lost to follow-up from each arm
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | FFR Guided PCI | CABG
Number analyzed (Participants) | 755 | 741
Participants
  Death | 12 | 7
  Death from cardiac causes | 6 | 4
Statistical Analysis 1: Comparison: FFR Guided PCI vs CABG; Test type: Other; Hazard Ratio (HR) = 1.7, 95% CI 2-sided [0.7 to 4.3]

5. Secondary Outcome: Number of Participants Experiencing Myocardial Infarction
Description: MI evaluated excluding patients lost to follow-up from each arm
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | FFR Guided PCI | CABG
Number analyzed (Participants) | 755 | 741
Participants
  Overall | 39 | 26
  Spontaneous | 25 | 17
  Procedural | 13 | 9
Statistical Analysis 1: Comparison: FFR Guided PCI vs CABG; Test type: Other; Hazard Ratio (HR) = 1.5, 95% CI 2-sided [0.9 to 2.5] — Hazard ratio for overall number of participants experiencing MI

6. Secondary Outcome: Number of Participants Experiencing Stroke
Description: Stroke evaluated excluding patients lost to follow-up from each arm.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | FFR Guided PCI | CABG
Number analyzed (Participants) | 755 | 741
Participants | 7 | 8
Statistical Analysis 1: Comparison: FFR Guided PCI vs CABG; Test type: Other; Hazard Ratio (HR) = 0.9, 95% CI 2-sided [0.3 to 2.4]

7. Secondary Outcome: Number of Participants Requiring Repeat Revascularization
Description: Any repeat revascularization evaluated excluding patients lost to follow-up from each arm
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | FFR Guided PCI | CABG
Number analyzed (Participants) | 755 | 741
Participants
  Overall | 45 | 29
  PCI | 39 | 26
  CABG | 6 | 3
Statistical Analysis 1: Comparison: FFR Guided PCI vs CABG; Test type: Other; Hazard Ratio (HR) = 1.5, 95% CI 2-sided [0.9 to 2.3] — Hazard ratio for overall number of participants experiencing repeat revascularization

8. Secondary Outcome: Number of Participants Experiencing BARC Type 3-5 Bleeding
Description: Bleeding Academic Research Consortium (BARC) type 3-5 indicates severe bleeding.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | FFR Guided PCI | CABG
Number analyzed (Participants) | 757 | 743
Participants | 12 | 28
Statistical Analysis 1: Comparison: FFR Guided PCI vs CABG; Test type: Other; p < 0.01, Fisher Exact

9. Secondary Outcome: Number of Participants Experiencing Acute Kidney Injury
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | FFR Guided PCI | CABG
Number analyzed (Participants) | 755 | 741
Participants | 1 | 7
Statistical Analysis 1: Comparison: FFR Guided PCI vs CABG; Test type: Other; p < 0.04, Fisher Exact

10. Secondary Outcome: Number of Participants Experiencing Atrial Fibrillation or Clinically Significant Arrhythmia
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | FFR Guided PCI | CABG
Number analyzed (Participants) | 757 | 743
Participants | 18 | 105
Statistical Analysis 1: Comparison: FFR Guided PCI vs CABG; Test type: Other; p < 0.001, Fisher Exact

11. Secondary Outcome: Number of Participants Experiencing Definite Stent Thrombosis
Time Frame: 1 year
Population: Outcome not assessed in CABG group (did not receive stent).
Measure: Count of Participants; unit: Participants
Arm/Group | FFR Guided PCI
Number analyzed (Participants) | 757
Participants | 6

12. Secondary Outcome: Number of Participants Experiencing Definite Symptomatic Graft Occlusion
Time Frame: 1 year
Population: Outcome not assessed in FFR guided PCI group (did not receive CABG).
Measure: Count of Participants; unit: Participants
Arm/Group | CABG
Number analyzed (Participants) | 743
Participants | 10

13. Secondary Outcome: Number of Participants Requiring Rehospitalization Within 30 Days
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | FFR Guided PCI | CABG
Number analyzed (Participants) | 757 | 743
Participants | 42 | 76
Statistical Analysis 1: Comparison: FFR Guided PCI vs CABG; Test type: Other; p < 0.001, Chi-squared

14. Secondary Outcome: MACCE
Description: Death, MI, stroke and any repeat revascularization (MACCE) rate at 2 years, 3 years and 5 years
Time Frame: 2 years, 3 years, 5 years
Reporting Status: Not Posted

15. Secondary Outcome: Death, MI, or Stroke at 5 Years
Description: Death, MI, or stroke at 5 years
Time Frame: 5 years
Reporting Status: Not Posted, anticipated posting 2025-05

16. Secondary Outcome: Individual Components of Primary Outcome
Description: Individual components of primary outcome: number of participants experiencing death, myocardial infarction, and stroke
Time Frame: At year 3
Population: FFR-guided PCI
Measure: Count of Participants; unit: Participants
Arm/Group | FFR Guided PCI | CABG
Number analyzed (Participants) | 757 | 743
Participants
  Death | 31 | 29
  Myocardial Infarction | 53 | 31
  Stroke | 12 | 15

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | FFR Guided PCI | CABG
All-Cause Mortality (participants affected / at risk) | 31/757 | 29/743
Serious Adverse Events (participants affected / at risk) | 91/757 | 68/743
Other Adverse Events (participants affected / at risk) | 45/757 | 29/743
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FFR Guided PCI (N=757) | CABG (N=743)
Death, MI or stroke (Cardiac disorders) | 91 | 68
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | FFR Guided PCI (N=757) | CABG (N=743)
Repeat revascularization (Cardiac disorders) | 45 | 29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-27): https://cdn.clinicaltrials.gov/large-docs/22/NCT02100722/Prot_SAP_000.pdf